CLINICAL TRIAL: NCT02161913
Title: Comparison of Two Psycho-educational Family Group Interventions for Persons With SCI and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Rehabilitation Institute (Other)
Collaborators: Washington State University (Other); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Douglas L. Weeks, Director of Research, St. Luke's Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHNF-288318
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCI Education Control Group (Active Comparator): The SCIEC condition is a 16-session, highly structured educational intervention that provides information on how SCI affects the body; methods for maximizing function, coping, and living with SCI; and staying healthy with SCI. It also includes general guidelines for improving health behavior. Each SCIEC session follows the same structure, beginning with a presentation of the objectives for the current session and a brief review of material from the previous session before introducing the session's topic and presenting information on one or two key problem areas. SCIEC utilizes a traditional didactic model with information delivered by an expert SCI educator in a classroom or lecture setting.
  Interventions: Behavioral: SCI Education Control Group
- Multi-family Group Treatment (Experimental): The MFG Program uses a structured problem-solving and skills training program to provide participants with SCI and their caregivers with tools and information to improve coping and help family members to connect through positive behavioral exchanges. MFG educators are health professionals with experience in management of SCI, such as physical therapists, recreational therapists, occupational therapists, and psychologists. MFG will last for 16 sessions across 9 months.
  Interventions: Behavioral: Multi-Family Group Treatment

INTERVENTIONS:
Behavioral: Multi-Family Group Treatment
  Arms: Multi-family Group Treatment
Behavioral: SCI Education Control Group
  Arms: SCI Education Control Group

SUMMARY:
Each year over 12,000 spinal cord injuries (SCI) occur in the United States. These injuries result in incredibly difficult, long-term, life adjustments both for patients and their caregivers. Many families continue to struggle with the physical, emotional and social impacts of SCI for months and years after the injury. Family education and support improves the outcomes of other challenging long-term conditions such as Traumatic Brain Injury, but little effort has been made to provide such interventions for persons with SCI and their caregivers. The proposed study will address this problem by refining and testing a group treatment for SCI called Multi-family Group (MFG) intervention. The groups will include people with SCI and their primary caregivers, and will be facilitated by an "educator" who is a health care provider who works with people with SCI. By providing education about the management of SCI and support in an MFG format, quality of life for persons with SCI is predicted to be improved. In turn, it is expected that caregivers will also benefit from the information, problem-solving activities, and social support that they receive from the educators and other group members. The investigators will recruit 32 individuals with SCI who have been discharged from inpatient rehabilitation within the previous three years and their primary caregivers. Participants will be randomized to the MFG intervention or to an education control condition and tested before and after treatment and 6 months following treatment. It is hypothesized that participants receiving MFG-SCI will have better outcomes than controls on measures of quality of life, health, and adjustment. The study will also test whether participants who are more recently discharged from inpatient rehabilitation will experience greater benefit from the MFG intervention or the education control intervention. If the outcomes support the hypotheses, the MFG intervention should be made available to those with SCI and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* For Person with SCI: quadriplegia or paraplegia due to an acquired injury with complete or incomplete lesion as defined by ASIA
* For person with SCI: discharge from inpatient rehabilitation within the previous 3 years
* For Person with SCI: age 18 years or older
* For Person with SCI: mobility impairment as the result of the SCI
* For Person with SCI: living in the community in a non-group setting after injury
* For Person with SCI: planning to remain in the geographic area for at least 12 months
* For Person with SCI: competency in English
* For Caregiver of Person with SCI: provision of instrumental or emotional support for a spouse, relative, partner, or friend with SCI for at least the past 6 months
* For Caregiver of Person with SCI: having regular contact with the individual with SCI (at least a minimum of 2 hours face-to-face contact per week)
* For Caregiver of Person with SCI: living with or near the individual with SCI
* For Caregiver of Person with SCI: over the age of 18
* For Caregiver of Person with SCI: having a telephone
* For Caregiver of Person with SCI: planning to remain in the geographic area for at least 12 months
* For Caregiver of Person with SCI: competency in English

Exclusion Criteria:

* For Person with SCI or Caregiver: terminal illness with life expectancy of less than 12 months
* For Person with SCI or Caregiver: in active treatment for cancer
* For Person with SCI or Caregiver: blind or deaf
* For Person with SCI or Caregiver: moderate to severe cognitive impairment (defined at screening as a score on the Short Portable Mental Status Questionnaire > 4 errors)
* For Person with SCI or Caregiver: severely high level of depression symptoms (defined at screening as a score on the CES-D >30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in ability to take action to improve one's health from baseline to end of treatment | 9 months
  Ability to take action to improve one's health will be assessed with the Patient Activation Measure (PAM) and the 8-item Short-Form Health Survey (SF-8). The PAM will measure the degree of individual's knowledge, confidence, and skill to participate in self-management. A higher degree of patient activation has been associated with better health outcomes for adults with chronic conditions. The SF-8 will assess self-reported general health, physical functioning, role-limitations due to physical health problems, bodily pain, and vitality.
Change in emotion regulation and interpersonal skills from baseline to end of treatment | 9 months
  Emotion regulation and interpersonal skills will be assessed with the Anger Expression Scale (AXS), the Abbreviated Duke Social Support Index (ADSSI), and the Family Crisis Oriented Personal Evaluation Scales (F-COPES). The AXS measures anger management including anger-in (suppression of angry feelings), anger-out (expression of anger towards property or people) and anger control (the frequency of attempts to control expressions of anger). The ADSSI measures both subjective support and social network interactions. The F-COPES assesses family-level coping including use of social/spiritual support, reframing negative events, and mobilizing the family to acquire/accept help.
Change in mental health and health behavior from baseline to end of treatment | 9 months
  Mental health and health behavior will be assessed for the presence and severity of depressive symptoms, substance use, and in caregivers, burden of care, as these may influence benefits derived from treatment. The 10-item Center for Epidemiologic Study of Depression (CESD-10) will measure depressive symptoms, and the Addiction Severity Index-Lite (ASI-L) will evaluate alcohol and substance use and related problems. The Caregiver Burden Inventory (CBI) will evaluate caregiver burden in four areas: physical, social, emotional and time dependence burden.

OTHER OUTCOMES:
Change in ability to take action to improve one's health from baseline to 6-months post-treatment | 15 months
  Ability to take action to improve one's health will be assessed with the Patient Activation Measure (PAM) and the 8-item Short-Form Health Survey (SF-8). The PAM will measure the degree of individual's knowledge, confidence, and skill to participate in self-management. A higher degree of patient activation has been associated with better health outcomes for adults with chronic conditions. The SF-8 will assess self-reported general health, physical functioning, role-limitations due to physical health problems, bodily pain, and vitality.
Change in emotion regulation and interpersonal skills from baseline to 6-months post-treatment | 15 months
  Emotion regulation and interpersonal skills will be assessed with the Anger Expression Scale (AXS), the Abbreviated Duke Social Support Index (ADSSI), and the Family Crisis Oriented Personal Evaluation Scales (F-COPES). The AXS measures anger management including anger-in (suppression of angry feelings), anger-out (expression of anger towards property or people) and anger control (the frequency of attempts to control expressions of anger). The ADSSI measures both subjective support and social network interactions. The F-COPES assesses family-level coping including use of social/spiritual support, reframing negative events, and mobilizing the family to acquire/accept help.
Change in mental health and health behavior from baseline to 6-months post-treatment | 15 months
  Mental health and health behavior will be assessed for the presence and severity of depressive symptoms, substance use, and in caregivers, burden of care, as these may influence benefits derived from treatment. The 10-item Center for Epidemiologic Study of Depression (CESD-10) will measure depressive symptoms, and the Addiction Severity Index-Lite (ASI-L) will evaluate alcohol and substance use and related problems. The Caregiver Burden Inventory (CBI) will evaluate caregiver burden in four areas: physical, social, emotional and time dependence burden.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G. Dyck, PhD, Principal Investigator — Washington State University; Douglas L. Weeks, PhD, Principal Investigator — St. Luke's Rehabilitation Institute
Locations (1):
- St. Luke's Rehabilitation Institute, Spokane, Washington, United States

REFERENCES:
- [Derived] Dyck DG, Weeks DL, Smith CL, Shaw M. Multiple family group intervention for spinal cord injury: Quantitative and qualitative comparison with standard education. J Spinal Cord Med. 2021 Jul;44(4):572-582. doi: 10.1080/10790268.2019.1710946. Epub 2020 Jan 21. PMID 31961284
- [Derived] Dyck DG, Weeks DL, Gross S, Lederhos Smith C, Lott HA, Wallace AJ, Wood SM. Comparison of two psycho-educational family group interventions for improving psycho-social outcomes in persons with spinal cord injury and their caregivers: a randomized-controlled trial of multi-family group intervention versus an active education control condition. BMC Psychol. 2016 Jul 26;4(1):40. doi: 10.1186/s40359-016-0145-0. PMID 27457478